CLINICAL TRIAL: NCT07279454
Title: The Eatwell Adapted Trial for Fibre Intervention in Bowel Cancer Risk Early-onset.
Brief Title: The EAT-FIBRE Study.
Acronym: EAT-FIBRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Cancer Research UK (Other); National Cancer Institute (NCI) (NIH); Bowelbabe Fund (Unknown); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 24/NW/0107
Record Dates: First submitted 2025-12-05; First posted 2025-12-12 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-11

CONDITIONS: Microbiome Related Mechanisms Linked to Early Onset Colorectal Cancer
Keywords: diet; fibre; EatWell; randomised controlled trial; microbiome; short-chain fatty acids; inflammation; twins
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EatWell diet (Active Comparator): Participants will be advised to follow the EatWell diet (UK national healthy eating guidance), providing 30g/day of dietary fibre.
  Interventions: Other: EatWell diet
- Modified EatWell diet (Experimental): Participants will be advised to follow the EatWell diet (UK national healthy eating guidance) with additional daily thresholds for fibre-rich food groups (wholegrain cereals, beans and pulses, and nuts and seeds), providing 40g/day of dietary fibre.
  Interventions: Other: Modified EatWell diet

INTERVENTIONS:
Other: Modified EatWell diet — 5-a-day for fruits and vegetables, <70g/day of red meat, 2 portions of fish/week (one of which is oily), <14 units of alcohol/week, plus specific daily thresholds of 180g/day (cooked) of wholegrain cereals, 160g/day (cooked) of beans and pulses, and 30g/day of nuts and seeds.
  Total dietary fibre = 40g/day.
  Arms: Modified EatWell diet
Other: EatWell diet — 5-a-day for fruits and vegetables, <70g/day of red meat, 2 portions of fish/week (one of which is oily), and <14 units of alcohol/week. No specific daily thresholds for wholegrain cereals, beans and pulses, or nuts and seeds will be provided.
  Total dietary fibre = 30g/day.
  Arms: EatWell diet

SUMMARY:
The goal of this clinical trial is to understand whether diet can impact mechanisms linked to early-onset colorectal cancer.

The main question it aims to answer is: does a high-fibre modified EatWell diet improve stool, blood, urine, and saliva measures linked to early-onset colorectal cancer, compared to the standard EatWell diet?

Researchers will compare the standard EatWell diet (UK national healthy eating guidance providing 30g/day of dietary fibre) to a modified EatWell diet (UK national healthy eating guidance plus specific thresholds for fibre-rich food groups providing 40g/day of dietary fibre).

Participants will follow the dietary advice for 12 weeks, attend clinic visits at the start and end of the study for stool, blood, urine, and saliva sampling, body composition measures, health checks, and complete health, diet, and lifestyle questionnaires.

DETAILED DESCRIPTION:
BACKGROUND The incidence of early-onset colorectal cancer (EOCRC) is on the rise worldwide. Many EOCRC cases may be preventable through modifiable lifestyle factors, including diet . Colorectal cancer risk reductions have been reported with higher intakes of dietary fibre, and different food sources of fibre may confer varying levels of protection. Dietary recommendations for colorectal cancer prevention advise limiting the intake of red and processed meats and added sugars, while prioritising fibre-rich foods such as fruits, vegetables, and whole grains, aligning with the UK EatWell diet; however, its effects on mechanisms underlying EOCRC remain to be elucidated.

AIM To evaluate whether a modified high-fibre EatWell diet can more effectively modulate metabolomic, microbiome, and inflammatory markers associated with EOCRC compared to the standard EatWell diet.

PARTICIPANTS One hundred adult twin pairs (n=200), volunteers of TwinsUK, will be invited to participate. Interested individuals will complete a screening survey and a food frequency questionnaire to determine eligibility.

METHODS EAT-FIBRE is a single-centre parallel-arm randomised controlled diet intervention trial. Twin pairs will be split-randomised with allocation to either the control arm (standard EatWell diet) or intervention arm (modified EatWell diet) to adhere to for 12 weeks. Participants will attend the clinic for stool, blood, urine, and saliva sampling, body composition measures, health checks, and complete health, diet, and lifestyle questionnaires, and will return at the endpoint for repeat measures. The follow-up will be remote at 12 months, where participants will collect and post stool, blood, urine, and saliva samples, and repeat various questionnaires.

ELIGIBILITY:
Inclusion

* If female, not pregnant, lactating, or planning a pregnancy within the next 4 months.
* Living in the United Kingdom.

Exclusion

* Dietary fibre intake <16 g/day or >30 g/day.
* Unwilling to comply with the intervention (wholegrains, beans and pulses, and nuts and seeds).
* Are diagnosed with the following food allergies: gluten, peanuts, or nuts.
* Are living or have a past medical history of an eating disorder.
* Alcohol Use Disorders Identification Test - Consumption score > 10 points.
* Have lost significant weight (>10% of original bodyweight) over the past 3 months.
* Use of any of the following drugs within the last month:

  (i) antifungals, antivirals, or antiparasitic medications (ii) methotrexate or immunosuppressive agents.
* Use of systemic antibiotics within the last 3 months.
* Use of commercial probiotics, prebiotics, laxatives, or other gut health supplements within the last month.
* Using Glucagon-Like Peptide-1 Receptor Agonists.
* Acute disease at the time of enrolment. Acute disease is defined as the presence of a moderate or severe illness with or without fever.
* Undergoing dietetic care for chronic conditions.
* History of cancer, except for squamous or basal cell carcinomas of the skin that have been medically managed by local excision.
* Any confirmed or suspected condition/state of immunosuppression or immunodeficiency (primary or acquired), including human immunodeficiency virus infection.
* Major surgery of the GI tract, except for cholecystectomy and appendectomy, in the past five years. Any major bowel resection at any time.
* Any other condition declared by the participant deemed by the medical supervisor to affect the normal conduct of the study and analysis of results.
* History of active, uncontrolled gastrointestinal disorders or diseases, including:

  (i) Coeliac disease (ii) inflammatory bowel disease, including ulcerative colitis, Crohn's disease, or indeterminate colitis (iii) persistent, infectious gastroenteritis, colitis or gastritis (iv) persistent or chronic diarrhoea of unknown aetiology (v) chronic constipation (vi) Irritable Bowel Syndrome (vii) Clostridium difficile infection (recurrent) (viii) Helicobacter pylori infection (untreated).
* Any other condition declared by the participant deemed by the medical supervisor to affect the normal conduct of the study and analysis of results.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Short Chain Fatty Acids | 12 weeks; from baseline to endpoint.
  Change from baseline in faecal butyrate.

SECONDARY OUTCOMES:
Microbially derived metabolites | 12 weeks; from baseline to endpoint.
  Change from baseline in faecal and circulating levels of microbially derived metabolites, including other SCFAs and bile acids.
Gut microbiome composition | 12 weeks; from baseline to endpoint.
  Change from baseline in faecal microbial community composition.
Markers of systemic and intestinal inflammation | 12 weeks; from baseline to endpoint.
  Change from baseline in circulating levels of inflammatory markers, including cytokines, and faecal levels of calprotectin and myeloperoxidase.

OTHER OUTCOMES:
Biomarkers of intestinal function | 12 weeks; from baseline to endpoint.
  Changes from baseline in markers of intestinal barrier function, including faecal levels of mucin-2 and circulating levels of intestinal fatty acid binding protein.
Prostaglandin E2 | 12 weeks; from baseline to endpoint.
  Change from baseline in urinary prostaglandin E2.
Markers of cardiometabolic health | 12 weeks; from baseline to endpoint.
  Change from baseline in circulating levels of individual markers related to cardiometabolic health, including glucose measured in mmol/L, and lipids measured in mmol/L.
Anthropometry | 12 weeks; from baseline to endpoint.
  Change from baseline in body composition, including weight in kilograms, height in meters for Body Mass Index (kg/m2) and adiposity measures, including % fat mass.

CONTACTS AND LOCATIONS:
Overall Officials: Jordana Bell, Professor, Principal Investigator — King's College London Twin Research & Genetic Epidemiology; Sarah Berry, Professor, Principal Investigator — King's College London Department of Nutritional Sciences
Locations (1):
- Department of Twin Research and Genetics, London, United Kingdom